CLINICAL TRIAL: NCT02337985
Title: Safety and Feasibility of Stem Cell Gene Transfer Following R-EPOCH for Non-Hodgkin Lymphoma in AIDS Patients Using Peripheral Blood Stem/Progenitor Cells Treated With a Lentivirus Vector-Encoding Multiple Anti-HIV RNAs
Brief Title: Gene Therapy and Combination Chemotherapy in Treating Patients With AIDS-Related Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14004; NCI-2014-02416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14004 (Other: City of Hope Medical Center); U01CA183012 (NIH)
Record Dates: First submitted 2014-12-23; First posted 2015-01-14 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: AIDS-Related Burkitt Lymphoma; AIDS-Related Diffuse Large B-cell Lymphoma; AIDS-Related Plasmablastic Lymphoma; AIDS-Related Primary Effusion Lymphoma; HIV Infection; AIDS Related Non-Hodgkin Lymphoma
MeSH Terms: conditions — HIV Infections | interventions — Prednisone; Rituximab; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (R-EPOCH, rHIV7-shI-TAR-CCR5RZ-transduced HSPC) (Experimental): Patients receive prednisone PO BID on days 1-5; rituximab IV on day 1; etoposide IV over 96 hours, doxorubicin hydrochloride IV over 96 hours and vincristine sulfate IV over 96 hours on days 1-4; and cyclophosphamide IV over 30-60 minutes on day 5. Patients then receive filgrastim SC QD beginning on day 6 and continuing until absolute neutrophil count recovers. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients then receive lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic stem/progenitor cells IV on day 0 (48 hours after the final combination chemotherapy course.)
  Interventions: Drug: Prednisone; Biological: Rituximab; Drug: Etoposide; Drug: Doxorubicin Hydrochloride; Drug: Vincristine Sulfate; Drug: Cyclophosphamide; Biological: Filgrastim; Biological: Lentivirus Vector rHIV7-shI-TAR-CCR5RZ-transduced Hematopoietic Stem/Progenitor Cells

INTERVENTIONS:
Drug: Prednisone — Given PO
Biological: Rituximab — Given IV
  Other Names: MOAB IDEC-C2B8
Drug: Etoposide — Given IV
  Other Names: Lastet; VP 16
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: Adriamycin
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Oncovin; VCR; Vincasar
Drug: Cyclophosphamide — Given IV
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Nivestim; r-metHuG-CSF; Neupogen
Biological: Lentivirus Vector rHIV7-shI-TAR-CCR5RZ-transduced Hematopoietic Stem/Progenitor Cells — Given IV
  Other Names: lentivirus-transduced hematopoietic progenitor cells

SUMMARY:
This pilot clinical trial studies gene therapy following combination chemotherapy in treating patients with acquired immune deficiency syndrome (AIDS)-related non-Hodgkin lymphoma. Placing genes that have been shown in the laboratory to inhibit the growth and spread of the immunodeficiency virus (HIV) into the patient's peripheral blood stem cells may improve the body's ability to fight HIV. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving gene therapy after combination chemotherapy may improve the body's ability to fight HIV and AIDS-related non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate the safety and feasibility of rHIV7-shI-TAR-CCR5RZ-treated hematopoietic stem progenitor cells (HSPC) (lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells) transplantation in AIDS patients completing treatment for non-Hodgkin lymphoma (NHL).

SECONDARY OBJECTIVES:

I. To determine the effect of HIV infection on the presence of gene-marked blood cells as measured by woodchuck post-transcriptional regulatory element (WPRE) deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) performed before, during, and after ATI.

II. To demonstrate the engraftment of gene-modified progeny cells following such treatment.

III. To determine if selection of these gene-modified progeny cells occurs during analytical treatment interruption (ATI) of combination anti-retroviral therapy (cART).

OUTLINE:

Patients receive prednisone orally (PO) twice daily (BID) on days 1-5; rituximab intravenously (IV) on day 1; etoposide, doxorubicin hydrochloride and vincristine sulfate IV over 96 hours on days 1-4; and cyclophosphamide IV over 30-60 minutes on day 5. Patients then receive filgrastim subcutaneously (SC) once daily (QD) beginning on day 6 and continuing until absolute neutrophil count recovers. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients then receive lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic stem/progenitor cells IV on day 0 (48 hours after the final combination chemotherapy course).

After completion of study treatment, patients are followed up at 1, 2, 3, 6, 9, 12, 18, and 24 months, every 6 months for 3 years, and then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive at or before the time of lymphoma diagnosis; all HIV positive patients are eligible regardless of HIV viral load or antiviral therapy (ART) status; all patients on study will receive ART as per standard guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Biopsy proven lymphoma for which rituximab, etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride (R-EPOCH) is appropriate frontline therapy, e.g., Burkitt lymphoma or diffuse large B-cell lymphoma (DLBCL) NHL, including plasmablastic lymphoma and primary effusion lymphoma but not T-cell lymphoma; tissue histology will be reviewed at the treating institution
* No psychosocial conditions that would hinder study compliance and follow-up
* Pretreatment serum glutamic oxaloacetic transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT) =< 2.5 x institutional upper limit of normal (ULN)
* Pretreatment serum bilirubin =< 2.5 x ULN or total bilirubin < 4.5 mg/dl with direct fraction =< 0.3 mg/dl in patients for whom these abnormalities are felt to be due to protease inhibitor therapy
* Patients with evidence of hepatitis C virus (HCV) or hepatitis B virus (HBV) infection must have no clinical evidence of cirrhosis
* Serum creatinine < 2 x the institutional ULN; however, if serum creatinine > 1.5 x ULN, a 24 hour urine creatinine clearance must be > 50 ml/min unless there is renal involvement by lymphoma
* Absence of clinically significant cardiomyopathy, congestive heart failure
* If the subject is female and of child bearing potential, subject must have negative serum or urine pregnancy test within 7 days of treatment with research agent; men with partners of child-bearing potential and women of child-bearing potential must be willing to use medically effective birth control methods, e.g. contraceptive pill, condom, or diaphragm and continue this for one year post HSPC infusion
* Subjects must be on a prophylactic regimen for Pneumocystis carinii pneumonia, or agree to begin such treatment and remain on treatment until after completion of therapy and until the cluster of differentiation (CD)4 cells are greater than 200/mm^3
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for 12 months following stem cell infusion; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent

ELIGIBILITY CRITERIA FOR HSPC TRANSPLANTATION

* Patients must demonstrate >= 75% disease reduction on computed tomography (CT) scan (confirmed by PET scan) after the third cycle of R-EPOCH relative to baseline, with no evidence of disease progression after the fifth cycle
* Subjects must complete the filgrastim (G-CSF)/plerixafor mobilization of peripheral blood progenitor cells, and subjects must have collected at least 5 x 10^6 CD34+ cells/kg by apheresis after Cycle 4

Exclusion Criteria:

* Any AIDS-related opportunistic infection occurring within the past year and for which treatment has been unsuccessful would be considered exclusionary, but this is done on a case-by-case basis as determined by the principal investigator (PI)
* Active cytomegalovirus (CMV) retinitis or other active CMV-related organ dysfunction; patients with a history of treated CMV infection are not excluded
* AIDS-related syndromes, infectious or otherwise, if perceived to cause excessive risk for morbidity post-HSPC infusion, as determined by the PI; examples include, but not limited to:

  * Severe AIDS-related wasting
  * Severe intractable diarrhea
  * Active inadequately treated opportunistic infection of the central nervous system (CNS)
  * Primary CNS lymphoma
* Pregnant or nursing women
* Any history of HIV-associated encephalopathy; dementia of any kind; seizures in the past 12 months
* Any perceived inability to directly provide informed consent (note: consent may not be obtained by means of a legal guardian)
* Any medical or physical contraindication or other inability to undergo HSPC collection
* Patients should not have any uncontrolled illness including ongoing or active infection other than HIV
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to G-CSF/filgrastim (E. coli producing cell line) and plerixafor
* Patients with other active malignancies; however, patients with skin cancers, namely basal cell or squamous cell carcinoma, and malignancies treated with curative intent having no known active disease present for >= 2 years, may be eligible
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-11-20 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events related to R-EPOCH, graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 2 years after completion of treatment
  Tables will be created to summarize these toxicities and side effects by dose and by course.
Incidence of adverse events related to lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic stem/progenitor cells infusion, graded using the NCI CTCAE version 4.03 | Up to 2 years
  All toxicities, related and unrelated, observed after each stem cell infusion will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI CTCAE and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Ability to obtain suitable numbers of lentiviral vector treated HSPC as determined by cell count | Up to day -2 (pre-infusion)
Presence of transgene in peripheral blood by digital droplet PCR | Up to 2 years

SECONDARY OUTCOMES:
Transgene ribonucleic acid expression by Northern blotting/hybridization and quantitative real-time PCR assay | Up to 15 years
HIV reservoir as determined by HIV-1 reverse transcriptase (RT)-PCR, DNA PCR, and DNA 2 long terminal repeat circle PCR | Up to 15 years and during ATI
HIV integration analysis by number of reads and loci | Up to 15 years
  Integration analyses will be done at month 6 and 12, and at week 16 of ATI, and at times when there is a clinical syndrome that suggests clonal expansion of hematopoietic cells.
Vector transgene sequences in peripheral blood mononuclear cells | Up to 2 years, possibly up to 15 years
Change in of shI-TAR-CCR5RZ-marked cells in bone marrow | Baseline to up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Krishnan, MD, Principal Investigator — City of Hope Medical Center; Mark J. Roschewski, MD, Principal Investigator — NCI Lymphoid Malignancy Branch
Locations (1):
- NCI Lymphoid Malignancies Branch, Bethesda, Maryland, United States